CLINICAL TRIAL: NCT05741437
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety After Oral Administration of CKD-378 and Co-administration of D745, D150 in Healthy Adults
Brief Title: A Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetics of CKD-378
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A129_01BE2225
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Type II Diabetes
Keywords: CKD-378
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: D745, D150 - A single oral dose of 2 tablets under food intake condition
  * Period 2: CKD-378 - A single oral dose of 1 tablet under food intake condition
  Interventions: Drug: CKD-378, QD, PO Drug: D745, D150, QD, PO
- Sequence 2 (Experimental): * Period 1: CKD-378 - A single oral dose of 1 tablet under food intake condition
  * Period 2: D745, D150 - A single oral dose of 2 tablets under food intake condition
  Interventions: Drug: CKD-378, QD, PO Drug: D745, D150, QD, PO

INTERVENTIONS:
Drug: CKD-378, QD, PO Drug: D745, D150, QD, PO — Durg: CKD-378, QD, PO Drug: D745, D150, QD, PO
  Other Names: CKD-378

SUMMARY:
A clinical trial to compare and evaluate the safety and pharmacokinetics of CKD-378

DETAILED DESCRIPTION:
A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety after Oral Administration of CKD-378 and Co-administration of D745, D150 in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged between 19 to 55 at screening
2. Weight ≥ 50kg(man) or 50kg(woman)
3. Body mass index (BMI) of 18.5 to 27.0kg/m2
4. If female, one of following conditions. Menopause (no menstruation more than 2 years) or surgically sterilized.
5. Those who agree to contraception from the first IP dosing day till 28 days after the last dosing day and decide not to provide sperm during the participation of clinical trial
6. Those who voluntarily decide to participate in paper and agree to comply with the cautions after fully understand the detailed description of this clinical trial

Exclusion Criteria:

1. Those who have clinically significant disease or medical history of Hepatopathy, Renal dysfunction, Neurological disorder, Immunity disorder, Respiratory disorder, Genitourinary system disorder, Haemato-oncology disorder, Cardiovascular disorder or Psychical disorder.
2. Those who are vulnerable to dehydration due to lack of ability in oral intake or have dehydration.
3. Those who had medical examination requiring radioactive iodine contrast material injected through IV 48 hours prior to first IP administration.
4. Those who have significant disease or medical history of urinary infection.
5. Those who have genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
6. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery which can interfere with drug absorption.
7. Those who have hypersensitivity to the main constituents or components of the investigational drug such as empagliflozin, metformin.
8. Those who have tested inappropriate in screening test 28 days prior to IP administration.

   * AST, ALT > 1.5 times higher than upper normal level
   * eGFR (estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
   * "Positive" or "Reactive" test result of Hepatitis B & C, HIV, RPR
   * Under 5 min resting condition, systolic blood pressure >150 mmHg or or <90 mmHg, diastolic blood pressure >100 mmHg or <50 mmHg.
9. Those who has a drug abuse history within one year or positive reaction on urine drug screening test.
10. Woman who are pregnant or breastfeeding
11. Those who exceed an alcohol, caffeine and cigarette consumption (caffeine> 5 cups/day, alcohol> 210g/week, smoking> 10 cigarettes/day) and not able to stop on smoking, caffeine and alcohol
12. Those who have used following drugs that can interfere with the study or have impact on safety of the subject.

    * ETC, herbal medicinal preparations within 14 days before the first dosing date
    * OTC, vitamins, health supplement within 7 days before the first dosing date
    * Depot injection or implantation within 30 days before the first dosing date
13. Those who received investigational products or participated in bioequivalence test within 180 days before the first administration of clinical trial drugs
14. Those who donated whole blood within 60 days before the first date of administration and donated ingredients within 30 days
15. Those who have received blood transfusion in 30 days
16. Those who are deemed insufficient to participate in clinical study by investigators

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
1. AUCt of CKD-378: Area under the concentration-time curve time zero to time | Pre-dose(0 hour) to 48 hours
2. Cmax of CKD-378: Maximum plasma concentration of the drug | Pre-dose(0 hour) to 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No